CLINICAL TRIAL: NCT02979366
Title: Phase I, International, Multicentre, Open-label, Non-randomised, Non-comparative Study of Intravenously Administered S64315, a Mcl-1 Inhibitor, in Patients With Acute Myeloid Leukaemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Phase I Study of S64315 Administred Intravenously in Patients With Acute Myeloid Leukaemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-64315-001; 2016-003768-38 (EudraCT Number); 136541 (Other: IND (FDA))
Record Dates: First submitted 2016-11-18; First posted 2016-12-01 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukaemia (AML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S64315 (also referred as MIK665) administered once a week (Experimental)
  Interventions: Drug: S64315 once a week
- S64315 (also referred as MIK665) administered twice a week (Experimental)
  Interventions: Drug: S64315 twice a week

INTERVENTIONS:
Drug: S64315 once a week — S64315 will be administered via i.v. infusion from 30 minutes and up to 3 hours once every week (21- day cycle), the starting dose is 50 mg. As data emerge during the study, the infusion duration and alternative dosing regimen may be changed.
  Other Names: MIK665
  Arms: S64315 (also referred as MIK665) administered once a week
Drug: S64315 twice a week — S64315 will be administered via i.v. infusion from 30 minutes and up to 3 hours twice every week (28- day cycle), the starting dose is 50 mg. As data emerge during the study, the infusion duration and alternative dosing regimen may be changed.
  Other Names: MIK665
  Arms: S64315 (also referred as MIK665) administered twice a week

SUMMARY:
The CL1-64315-001 study is a phase I, international, multicentre, open-label, non-randomised, non-comparative study. This study is designed in two parts: one part for dose escalation, one part for dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years;
* Patients with cytologically confirmed and documented de novo, secondary or therapy-related AML, excluding acute promyelocytic leukaemia (APL, French-American British M3 classification):

  * with relapsed or refractory disease without established alternative therapy or
  * secondary to MDS treated at least by hypomethylating agent or
  * > 65 years not previously treated for AML and who are not candidates for intensive chemotherapy nor candidates for established alternative chemotherapy Or Patients with cytologically confirmed and documented MDS), in relapse or refractory after previous treatment line including at least one hypomethylating agent and have ≥10% bone marrow blasts;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Circulating white blood cells < 10^9 /L (with or without use of hydroxycarbamide).
* Adequate renal function defined as:

  • Serum creatinine ≤ 1.5 x ULN (upper normal limit) or calculated creatinine clearance (determined by MDRD) > 50 mL/min/1.73m2.
* LDH < 2 x ULN
* Adequate hepatic function defined as:

  * AST and ALT ≤ 1.5 x ULN
  * Total bilirubin level ≤ 1.5 x ULN, except for patients with known Gilbert's syndrome (confirmed by the UGT1A1 polymorphism analysis), who are excluded if total bilirubin>3.0 x ULN or direct bilirubin > 1.5 x ULN
* Serum CK/CPK ≤2.5 x ULN.

Exclusion Criteria:

* Unlikely to cooperate in the study.
* Participant already enrolled in the study who has received at least one S64315 infusion.
* Pregnancy, breastfeeding or possibility of becoming pregnant during the study.
* Participation in another interventional study requiring investigational treatment intake within 2 weeks or at least 5 half-lives (whichever is longer) prior to first dose of S64315 (participation in non-interventional registries or epidemiological studies is allowed).
* Presence of ≥ CTCAE grade 2 toxicity (except alopecia of any grade) due to prior cancer therapy, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 4.03)
* Unresolved ≥ CTCAE grade 2 diarrhoea or medical conditions associated with chronic diarrhoea (such as irritable bowel syndrome, inflammatory bowel disease)
* Known carriers of HIV antibodies
* Known history of significant liver disease
* Uncontrolled hepatitis B or C infection
* Known active or chronic pancreatitis
* History of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG) within 6 months prior to starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs during the first cycle of treatment with single agent S64315 | 21-day cycle 1
Safety tolerance profile of S64315 assessed by:Incidence and severity of AEs | From first dose until 30 days after the last dose administration
Tolerability: Dose interruptions | From first dose until 30 days after the last dose administration
Tolerability: Dose reductions | From first dose until 30 days after the last dose administration
Tolerability: Dose intensity | From first dose until 30 days after the last dose administration

SECONDARY OUTCOMES:
Concentration at the end of infusion (C inf) in plasma | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Cumulative amount of a compound excreted in the urine (Ae) | only D1 of cycle 1
Preliminary efficacy assessment according to Cheson criteria (adapted for each disease) | From first dose until 30 days after the last dose administration
Time corresponding to end of infusion (tinf/tend) in plasma | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Area under the concentration-time curve from zero (time of drug administration) to tlast (AUC last) in plasma | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Time corresponding to Clast (tlast) in plasma. | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Last quantifiable observed concentration (Clast) in plasma | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Area Under the Curve (AUC) in plasma | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Terminal elimination half-life (t½,z) in plasma | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
total Clearance (CL) | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Volume of distribution at steady-state (Vss) in plasma | D1 and D2 of cycle 1 and 2, D15 and D16 of cycle 1 and D1 from cycle 3 to cycle 6.
Ae expressed as a percentage of the dose (fe) in urine | only D1 of cycle 1
Renal clearance (CLR) | only D1 of cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Andrew WEI, Principal Investigator — The Alfred Hospital, Melbourne, Victoria
Locations (9):
- United States (2):
  - Patient Care Location: Smilow Cancer Hospital at Yale, New Haven, Connecticut
  - The University of Texas MD Anderson Cancer Center, Department of Leukemia, Division of Cancer Medicine, Houston, Texas
- Australia (2):
  - The Alfred Hospital Department of Haematology, Melbourne
  - Royal Melbourne Hospital, Department of Clinical Haematology and BMT Service, Melbourne
- France (3):
  - Institut Paoli-Calmettes Departement d'Hématologie, Marseille
  - Hôpital Saint-Antoine Département d'Hematologie Clinique et de Thérapie cellulaire, Paris
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
- Spain (2):
  - Hospital Universitario Vall d' Hebron/VHIO Hematology Department, Barcelona
  - Hospital Universitario La Fe Hematology Department, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com

REFERENCES:
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/